CLINICAL TRIAL: NCT04161872
Title: Evaluation of the Effects of a Supplement Composed by Quercetin, Rutin, Bromelain and L-carnosine in Patients With Hyperuricemia, a Randomized Clinical Trial
Brief Title: Nutraceutical on Hyperuricemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-20180016368
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uricemin (Active Comparator)
  Interventions: Drug: Uricemin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Uricemin — Uricemin is a nutraceutical containing quercetin, rutin, bromelain and L-carnosine
  Arms: Uricemin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this study will be to evaluate if a nutraceutical containing quercetin, rutin, bromelain and L-carnosine (Uricemin®) can reduce uric acid levels in subjects with values between ≥ 6 and < 7 mg/dl after 3 months of therapy.

DETAILED DESCRIPTION:
The aim of this study will be to evaluate if a nutraceutical containing quercetin, rutin, bromelain and L-carnosine (Uricemin®) can reduce uric acid levels in subjects with values between ≥ 6 and < 7 mg/dl after 3 months of therapy.

Patients will be randomized to Uricemin® or placebo for three months. We will evaluate body weight, fasting plasma glucose (FPG), lipid profile, uricemia (UA), high-sensitivity C-reactive protein (Hs-CRP) at baseline and after 3 months since the study start. Treatment tolerability will be assessed evaluating transaminases, and creatinine, and all adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uric acid levels between ≥ 6 and < 7 mg/dl
* Patients not taking hypouricemic agents (both pharmaceuticals or nutraceutical agents)

Exclusion Criteria:

* Patients with previous gout attack
* Patients with impaired hepatic function
* Patient with impaired renal function
* Patients with gastrointestinal disorders
* Patients with current or previous evidence of ischemic heart disease, heart failure, or stroke
* Patients with weight change of > 3 Kg during the preceding 3 months
* Patients with history of malignancy, and significant neurological or psychiatric disturbances, including alcohol or drug abuse.
* Patients taking (within the previous 3 months) hypouricemic agents, laxatives, beta-agonists (other than inhalers), cyproheptadine, antidepressants, antiserotoninergics, phenothiazines, barbiturates, oral corticosteroids, and antipsychotics
* Women who were pregnant or breastfeeding or of childbearing potential and not taking adequate contraceptive precautions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Variation of Hyperuricemia | 3 months
  Uric acid levels

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy